CLINICAL TRIAL: NCT02976714
Title: Identification of Predictive Epigenetic Biomarkers of Lung Disease Severity in Cystic Fibrosis
Acronym: MethylBiomark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL16_0256
Record Dates: First submitted 2016-11-08; First posted 2016-11-29 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Lung disease; DNA methylation; Predictive biomarkers
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CF patients (Other): CF patients carry a spontaneous sputum that is made in the context of bronchial drainage sessions conducted as part of usual care.
  Interventions: Other: spontaneous sputum

INTERVENTIONS:
Other: spontaneous sputum — CF patients carry a spontaneous sputum that is made in the context of bronchial drainage sessions conducted as part of usual care (inclusion, 6 months, 12 months, 18 months).
  The collection of spontaneous sputum is carried out within the bronchial drainage sessions, which are routinely performed at each visit. The spontaneous sputum is collected in a sterile container. In order not to contaminate the sputum with buccal epithelial cells will be asked patients to rinse the mouth before expectorate.

SUMMARY:
The general aims of this project are (i) to identify predictive epigenetic biomarkers of lung disease severity in Cystic Fibrosis, (ii) to characterize a non-invasive cellular model, spontaneous sputum, for the analysis of these epigenetic biomarkers, (iii) to analyze the variations in DNA methylation for a same patient over time.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is an autosomal recessive disease resulting from mutations in the CFTR gene. CFTR encodes a chloride channel, mainly expressed at the apical membrane of epithelial cells. CFTR dysfunction induces mucus thickening, causing multiple disorders in respiratory, digestive and reproductive tracts. In CF patients, lung disease is the main cause of morbidity and mortality, and its severity is variable among CF patients, even among those with the same genotype. This clinical variability depends on two factors: genetic (complex alleles of CFTR gene and modifier genes) and environmental factors. Genetic factors have been largely explored, and several modifier genes have been identified. By contrast, environmental factors are still poorly known. It is well established that environmental factors modify the phenotype by acting on epigenetic marks (i.e. DNA methylation, histone modification) present in the genome. Epigenetic modifications regulate and modulate gene expression.

In a previous we profiled DNA methylation genome-wide in nasal epithelial cell samples from 32 CF patients and 24 healthy controls. CF patients homozygous for the p.Phe508del mutation and >18-years-old were stratified according to the lung disease severity. Through this study, we identified 187 genomic regions (CpG dinucleotides) differentially methylated between CF patients with mild lung disease and CF patients with severe lung disease. The present project aims at identifying predictive epigenetic biomarkers of lung disease severity, among these 187 regions. While the previous study was carried out on genomic DNA extracted from nasal epithelial cells, in the present project we will use a non-invasive model: spontaneous sputum.

Hypothesis: some differentially methylated genomic regions between mild and severe CF patients can be used as predictive epigenetic biomarkers of lung disease severity in cystic fibrosis.

Objectives: (i) to identify predictive epigenetic biomarkers of lung disease severity among the differentially methylated genomic regions between mild and severe CF patients, (ii) to characterize a non-invasive cellular model, spontaneous sputum, for the analysis of epigenetic biomarkers of lung disease severity in CF, (iii) to analyze the variations in DNA methylation for a same patient over time (at time of inclusion, 6 months, 12 months and 18 months)

ELIGIBILITY:
Inclusion Criteria:

* free and informed consent obtained, and consent signed
* subject covered by a state insurance scheme
* women and men aged 12 to 30
* subject affected by cystic fibrosis, carrier of two severe mutations in trans (in the same allele) in the CFTR gene
* subject able to realize a spirometry before and during the study

Exclusion Criteria:

* subject in an exclusion period of a previous study
* subject placed under judicial protection, guardianship or supervision
* impossibility to give informed information to the subject
* subject who does not read fluently French
* pregnancy
* breastfeeding
* transplanted subject

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
DNA methylation | at time of inclusion
  Spontaneous expectoration at baseline
DNA methylation | 6 months
  Spontaneous expectoration at 6 months
DNA methylation | 12 months
  Spontaneous expectoration at 12 months
DNA methylation | 18 months
  Spontaneous expectoration at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided